CLINICAL TRIAL: NCT00957697
Title: Pain After Stroke, Part 2: Clinical Characteristics and Classification of Pain in Patients After Stroke
Status: Completed | Type: Observational
Sponsor: Danish Pain Research Center (Other)
Responsible Party: Sponsor
Other Study IDs: 20060083
Record Dates: First submitted 2009-08-11; First posted 2009-08-12 (Estimated); Last update posted 2011-08-30 (Estimated); Status verified 2011-08

CONDITIONS: Pain
Keywords: Central Neuropathic Pain; Central Post-Stroke Pain; Stroke; Pain
MeSH Terms: conditions — Pain; Stroke

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No

SUMMARY:
The purpose of this study is to investigate the prevalence of characteristics of pain in a cohort of patients with prior stroke suspected of having central post stroke pain, identified through a postal questionnaire.

DETAILED DESCRIPTION:
Medical history, pain history, pain drawing, DN4, sensory examination.

ELIGIBILITY:
Inclusion Criteria:

* Possible neuropathic pain following stroke

Exclusion Criteria:

* Severe dementia
* Severe language barriers
* Patients who cannot cooperate

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Cohort of stroke patients diagnosed in 2004-2005 in the County of Aarhus identified through the National Indicator Project Stroke Database of Denmark
Sampling Method: Non-Probability Sample
Enrollment: 52 (Actual)
Dates: Start 2008-04; Primary Completion 2010-05 (Actual); Study Completion 2010-07 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Henriette Klit, MD, Principal Investigator — Danish Pain Research Center